CLINICAL TRIAL: NCT03309410
Title: Is Mathematical Arterialized Peripheral Venous Blood Gas Reliable Compared to Arterial Blood Gas? - a Clinical Validation Study
Brief Title: Mathematical Arterialization of Venous Blood Gas
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Department of Anesthesiology, North Denmark Regional Hospital (Unknown); Center for Clinical Research, North Denmark Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Mads Lumholdt, Principal investigator, Aalborg University
Other Study IDs: vTAC-Pilot
Record Dates: First submitted 2017-10-05; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Matched-Pair Analysis; Blood Gas Analysis; Emergency Service, Hospital
Keywords: Blood Gas Analysis; Emergency Service, Hospital; Venous to arterial conversion; Matched-Pair Analysis
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-study: In the pre-study, venous samples were collected in paired 2 mL ABG syringes and 4.5 mL tubes from each of the 10 patients, to determine which blood collection method was preferred. VBG samples were collected via a butterfly needle with a three-way stopcock in conjunction with routine venous blood sampling upon admission. VBG samples were collected by the biomedical laboratory technician in the same manner as PVB samples in the normal clinical setting. Results from the pre-study were used to determine the preferred blood collection method in the main study. In this study, paired ABG and VBG samples were collected simultaneously from each of the 20 patients. The ABG samples were collected by the responsible physician. Allocation to either the pre-study or the main study was performed by simple quasi-random allocation in order of admission.
  Interventions: Diagnostic Test: Venous to arterial conversion (v-TAC)
- Main study: In this study, paired ABG and VBG samples were collected simultaneously from each of the 20 patients. The ABG samples were collected by the responsible physician. Allocation to either the pre-study or the main study was performed by simple quasi-random allocation in order of admission. The clinical indication for ABG analysis was decided by the responsible physician in the ED upon patient admission and based on national guidelines and criteria.
  Interventions: Diagnostic Test: Venous to arterial conversion (v-TAC)

INTERVENTIONS:
Diagnostic Test: Venous to arterial conversion (v-TAC) — This was an observational study. Paired arterial blood gas and venous blood gas was drawn from each patient and compared. Venous blood gas was converted to arterial blood gas values using v-TAC.

SUMMARY:
Objective: Arterial blood gas (ABG) analysis is essential in the clinical assessment of potential acutely ill patients. Venous to arterial conversion (v-TAC), a mathematical method, has recently been developed to convert peripheral venous blood gas (VBG) values to arterialized VBG (aVBG) values. The aim of this study was to test the reliability of aVBG compared to ABG in an emergency department (ED) setting.

Method: Twenty ED patients were included in this study. ABG and three aVBG samples were collected from each patient. The aVBG samples were processed in three different ways for comparison: aVBG1 was held steady and analysed within 5 minutes; aVBG2 was tilted in 5 minutes and analysed within 7 minutes; aVBG3 was held steady and analysed after 15 minutes. All VBG samples were arterialized using the v-TAC method. ABG and aVBG samples were compared using Lin's Concordance Correlation Coefficient (CCC) and Bland-Altman's analysis.

DETAILED DESCRIPTION:
Arterial blood gas (ABG) analysis is essential in assessment of respiratory and metabolic status in acutely ill patients. In comparison to peripheral venous blood (PVG) sampling, the ABG sampling procedure is more painful for the patient and technically more challenging for the clinician to perform. Other drawbacks of ABG sampling include adverse events such as subcutaneous hematoma, arterial thrombosis or embolization, and the serious, though rare, complication pseudoaneurysms.

Peripheral venous blood gas (VBG) sampling has been suggested as an alternative to the ABG procedure. This procedure causes less patient discomfort and the sample can be analysed in combination with other venous blood tests. Studies have revealed that pH and bicarbonate have good correlation, whereas venous and arterial blood gasses (pO2 and pCO2) show low agreement. A recent systematic review comparing ABG and VBG in the ED setting found similar results and concluded that venous pCO2 was not an accurate representative of arterial pCO2.

However, a new method has been developed to calculate ABG values mathematically from peripheral venous blood by use of venous to arterial conversion (v-TAC) software (Obimedical, Denmark), supplemented with oxygen saturation measured by pulse oximetry. The principle of the method is a mathematical transformation of VBG values to arterialized values (aVBG) by simulating the transport of blood back through the tissue. To facilitate this simulation the following physiologically relevant assumptions were made: 1) The peripheral extremity was well perfused; 2) change in base excess across the tissue sampling site was approximately zero; 3) the respiratory quotient (rate of CO2 production and O2 utilisation over capillaries) could not vary outside the range 0.7 and 1.0, and 4) the haemoglobin concentration was constant from artery to vein. Initial testing of the method in an emergency department setting showed acceptable clinical congruence between arterial and mathematically arterialized pH and pCO2 with a small difference on 0.001- 0.024 and 0.00 0.46 kPa, respectively. However, inaccurate values of pO2 were seen when oxygen saturation measured by pulse oximetry was above 96%, due to the flat shape of the oxygen dissociation curve (ODC).

The aim of this study was to test appropriate practical handling of venous blood gas samples and evaluate the reliability of the v-TAC method, in an acute medical emergency setting in awake and circulatory stable patients capable of giving consent.

Methods Patient inclusion The study was conducted in the ED at North Denmark Regional Hospital from September through October 2015 in daytime. This hospital is 24-hour hospital with a collective medical and abdominal surgery emergency department, with 7-10.000 annual admissions per year.

Circulatory stable patients needing ABG analysis for respiratory and metabolic assessment were selected randomly for participation in the study. Patients were considered circulatory stable if systolic blood pressure was above 90 mmHg and heart rate was 50 to 110 beats/min in accordance with Danish Emergency Process Triage (DEPT), which were used to triage patients upon admission. A total of 30 patients were included; 10 patients for a pre-study purpose and then 20 patients in the following main study. Allocation to either the pre-study or the main study was performed by simple quasi-random allocation in order of admission. The clinical indication for ABG analysis was decided by the responsible physician in the ED upon patient admission and based on national guidelines and criteria.

Blood collection In the pre-study, venous samples were collected in paired 2 mL ABG syringes and 4.5 mL tubes from each of the 10 patients, to determine which blood collection method was preferred. VBG samples were collected via a butterfly needle with a three-way stopcock in conjunction with routine venous blood sampling upon admission. VBG samples were collected by the biomedical laboratory technician in the same manner as PVB samples in the normal clinical setting. Results from the pre-study were used to determine the preferred blood collection method in the main study. In this study, paired ABG and VBG samples were collected simultaneously from each of the 20 patients. The ABG samples were collected by the responsible physician.

Blood analysis Blood for VBG analysis collected in the syringe and 4.5 mL tube in the pre-study were analysed within five minutes after sampling. In the main study blood for VBG analysis was collected in three 4.5 mL tubes and converted to arterialised VBG (referred to as aVBG). Each aVBG tube was processed differently as follows: aVBG1 was held steady and analysed within five minutes of sample collection, aVBG2 was tilted in five minutes and analysed after seven minutes and aVBG3 was handled as aVBG1, but analysed after fifteen minutes. ABG samples were analysed within five minutes after sampling. All ABG and VBG samples were analysed with ABL800 blood gas analyser (Radiometer, Denmark) an VBG samples were mathematically converted to aVBG using v-TAC software which was integrated into the ABL800 analyser. In our hospital, the reference values for ABG parameters are as follows: pH 7.37-7.45, pCO2 4.30-6.00 kPa, and pO2 9.60-14.4 kPa. All results from analysed ABG and aVBG samples were registered automatically in the hospital database. On the standard of care basis, only the ABG results were used as the usual standard reference in the medical evaluation of the patients, who took part in the study.

Ethics and data protection The Danish Research Ethics Committee in the North Denmark Region was notified. Since the v-TAC method has previously been approved to be used in clinical research and blood sampling was performed as routine practice, ethical approval was not required. This study was approved by the Danish Data Protection Agency.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the emergency department.
* Need for ABG for respiratory or metabolic assessment.

Exclusion Criteria:

* Circulatory unstable patients (systolic blood pressure < 90mmHg og heart rate <50beats/min or >110beats/min).

Age Groups: Child, Adult, Older Adult
Study Population: Circulatory stable patients needing ABG analysis for respiratory and metabolic assessment were selected randomly for participation in the study. Patients were considered circulatory stable if systolic blood pressure was above 90 mmHg and heart rate was 50 to 110 beats/min in accordance with Danish Emergency Process Triage (DEPT), which were used to triage patients upon admission. A total of 30 patients were included; 10 patients for a pre-study purpose and then 20 patients in the following main study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Lin's Concordance correlation coefficient | 1 day
  Comparison of venous pH between glass and syringe samples.
Lin's Concordance correlation coefficient | 1 day
  Comparison of venous pCO2 (Unit of Measurement: kilopascal) between glass and syringe samples.
Lin's Concordance correlation coefficient | 1 day
  Comparison of venous pO2 (Unit of Measurement: kilopascal) between glass and syringe samples.
Bland and Altman plot | 1 day
  Comparison of venous pH between glass and syringe samples.
Bland and Altman plot | 1 day
  Comparison of venous pCO2 (Unit of Measurement: kilopascal) between glass and syringe samples.
Bland and Altman plot | 1 day
  Comparison of venous pO2 (Unit of Measurement: kilopascal) between glass and syringe samples.
Lin's Concordance correlation coefficient | 1 day
  Comparison of pH between aVBG and ABG.
Lin's Concordance correlation coefficient | 1 day
  Comparison of pCO2 (Unit of Measurement: kilopascal) between aVBG and ABG.
Lin's Concordance correlation coefficient | 1 day
  Comparison of pO2 (Unit of Measurement: kilopascal) between aVBG and ABG.
Bland and Altman plot | 1 day
  Comparison of pH between aVBG and ABG.
Bland and Altman plot | 1 day
  Comparison of pCO2 (Unit of Measurement: kilopascal) between aVBG and ABG.
Bland and Altman plot | 1 day
  Comparison of pO2 (Unit of Measurement: kilopascal) between aVBG and ABG.

SECONDARY OUTCOMES:
Hemoglobin concentration | 1 day
  Comparison of venous blood hemoglobin (Unit of Measurement: mmol/L) between glass and syringe blood.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Christensen, Study Chair — Aalborg University; Peter Leutscher, Study Director — Center for Clinical Research, North Denmark Regional Hospital

IPD SHARING:
Plan to Share IPD: No
Sensitive individual participant data (IPD) will not be available to other researchers. IPD will be kept in a secure personal drive within the regions server. All sensitive IPD will be anonymized before publication.

REFERENCES:
- [Background] Dar K, Williams T, Aitken R, Woods KL, Fletcher S. Arterial versus capillary sampling for analysing blood gas pressures. BMJ. 1995 Jan 7;310(6971):24-5. doi: 10.1136/bmj.310.6971.24. No abstract available. PMID 7827548
- [Background] Matheson L, Stephenson M, Huber B. Reducing pain associated with arterial punctures for blood gas analysis. Pain Manag Nurs. 2014 Sep;15(3):619-24. doi: 10.1016/j.pmn.2013.06.001. Epub 2014 Feb 24. PMID 24572291
- [Background] Leone V, Misuri D, Console N. Radial artery pseudoaneurysm after a single arterial puncture for blood-gas analysis: a case report. Cases J. 2009 Jul 21;2:6890. doi: 10.4076/1757-1626-2-6890. PMID 19829877
- [Background] Dev SP, Hillmer MD, Ferri M. Videos in clinical medicine. Arterial puncture for blood gas analysis. N Engl J Med. 2011 Feb 3;364(5):e7. doi: 10.1056/NEJMvcm0803851. No abstract available. PMID 21288091
- [Background] Zavorsky GS, Cao J, Mayo NE, Gabbay R, Murias JM. Arterial versus capillary blood gases: a meta-analysis. Respir Physiol Neurobiol. 2007 Mar 15;155(3):268-79. doi: 10.1016/j.resp.2006.07.002. Epub 2006 Aug 17. PMID 16919507
- [Background] Ak A, Ogun CO, Bayir A, Kayis SA, Koylu R. Prediction of arterial blood gas values from venous blood gas values in patients with acute exacerbation of chronic obstructive pulmonary disease. Tohoku J Exp Med. 2006 Dec;210(4):285-90. doi: 10.1620/tjem.210.285. PMID 17146193
- [Background] McCanny P, Bennett K, Staunton P, McMahon G. Venous vs arterial blood gases in the assessment of patients presenting with an exacerbation of chronic obstructive pulmonary disease. Am J Emerg Med. 2012 Jul;30(6):896-900. doi: 10.1016/j.ajem.2011.06.011. Epub 2011 Sep 9. PMID 21908141
- [Background] Kelly AM. Can VBG analysis replace ABG analysis in emergency care? Emerg Med J. 2016 Feb;33(2):152-4. doi: 10.1136/emermed-2014-204326. Epub 2014 Dec 31. PMID 25552544
- [Background] Bloom BM, Grundlingh J, Bestwick JP, Harris T. The role of venous blood gas in the emergency department: a systematic review and meta-analysis. Eur J Emerg Med. 2014 Apr;21(2):81-8. doi: 10.1097/MEJ.0b013e32836437cf. PMID 23903783
- [Background] Rees SE, Toftegaard M, Andreassen S. A method for calculation of arterial acid-base and blood gas status from measurements in the peripheral venous blood. Comput Methods Programs Biomed. 2006 Jan;81(1):18-25. doi: 10.1016/j.cmpb.2005.10.003. Epub 2005 Nov 21. PMID 16303205
- [Background] Tygesen G, Matzen H, Gronkjaer K, Uhrenfeldt L, Andreassen S, Gaardboe O, Rees SE. Mathematical arterialization of venous blood in emergency medicine patients. Eur J Emerg Med. 2012 Dec;19(6):363-72. doi: 10.1097/MEJ.0b013e32834de4c6. PMID 22082876
- [Background] Skriver C, Lauritzen MM, Forberg JL, Gaardboe-Poulsen OB, Mogensen CB, Hansen CL, Berlac PA. [Triage quickens the treatment of the most sick patients]. Ugeskr Laeger. 2011 Oct 3;173(40):2490-3. Danish. PMID 21975184
- [Background] Toftegaard M, Rees SE, Andreassen S. Evaluation of a method for converting venous values of acid-base and oxygenation status to arterial values. Emerg Med J. 2009 Apr;26(4):268-72. doi: 10.1136/emj.2007.052571. PMID 19307387
- [Background] Collins JA, Rudenski A, Gibson J, Howard L, O'Driscoll R. Relating oxygen partial pressure, saturation and content: the haemoglobin-oxygen dissociation curve. Breathe (Sheff). 2015 Sep;11(3):194-201. doi: 10.1183/20734735.001415. PMID 26632351
- [Background] Kelly AM, McAlpine R, Kyle E. Venous pH can safely replace arterial pH in the initial evaluation of patients in the emergency department. Emerg Med J. 2001 Sep;18(5):340-2. doi: 10.1136/emj.18.5.340. PMID 11559602
- [Background] Ibrahim I, Ooi SB, Yiong Huak C, Sethi S. Point-of-care bedside gas analyzer: limited use of venous pCO2 in emergency patients. J Emerg Med. 2011 Aug;41(2):117-23. doi: 10.1016/j.jemermed.2008.04.014. Epub 2008 Oct 18. PMID 18930370
- [Background] Hedberg P, Majava A, Kiviluoma K, Ohtonen P. Potential preanalytical errors in whole-blood analysis: effect of syringe sample volume on blood gas, electrolyte and lactate values. Scand J Clin Lab Invest. 2009;69(5):585-91. doi: 10.1080/00365510902878716. PMID 19396657
- [Background] Castagneto M, Giovannini I, Boldrini G, Nanni G, Pittiruti M, Sganga G, Castiglioni GC. Cardiorespiratory and metabolic adequacy and their relation to survival in sepsis. Circ Shock. 1983;11(2):113-30. PMID 6416705
- [Background] Lauscher P, Lauscher S, Kertscho H, Habler O, Meier J. Hyperoxia reversibly alters oxygen consumption and metabolism. ScientificWorldJournal. 2012;2012:410321. doi: 10.1100/2012/410321. Epub 2012 May 1. PMID 22623894
- See also: Arteriepunktur - Lægehåndbogen (Arterial Blood Gas - Doctor's Handbook) — https://www.sundhed.dk/sundhedsfaglig/laegehaandbogen/undersoegelser-og-proever/kliniske-procedurer/hjertekar/arteriepunktur/